CLINICAL TRIAL: NCT05400941
Title: Adapting and Implementing Evidence-based Breast Cancer Follow-up in Primary Care
Brief Title: Aim 3, Adapting and Implementing Evidence-based Breast Cancer Follow-up in Primary Care
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Shawna V. Hudson, PhD, Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro2021000838; R01CA257197 (NIH)
Record Dates: First submitted 2022-05-23; First posted 2022-06-02 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2024-11

CONDITIONS: Cancer, Breast; Health Care Utilization
MeSH Terms: conditions — Breast Neoplasms; Patient Acceptance of Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Practice Led Intervention (Active Comparator): Clinic staff will participate in learning collaborative and practice facilitation as well as receive expert consultation and audit and feedback.
  Interventions: Behavioral: Practice Led Intervention
- Standard of Care (No Intervention): No intervention.

INTERVENTIONS:
Behavioral: Practice Led Intervention — This is a quality improvement intervention that includes learning collaboratives, practice facilitation, expert consultation and audit and feedback.
  Arms: Practice Led Intervention

SUMMARY:
This mixed methods study evaluates the effectiveness of an organizational intervention to enhance implementation of strategies to increase breast cancer survivorship symptom and risk management.

DETAILED DESCRIPTION:
Aim 3 is a hybrid type 1 effectiveness-implementation cluster randomized study with a waitlist control in 26 primary care practices. This study uses a tailored combination of practice facilitation, expert consultation, collaborative learning events, and audit and feedback as intervention strategies, and a mixed-methods comparative case study learning evaluation for primary care practices to adapt priority recommendations of evidence-based activities for breast cancer survivorship care. Intervention effectiveness will be assessed in two groups of clinics: 13 cases that will receive the implementation intervention and 13 waitlist controls. Impact of this implementation will be measured using mixed methods to assess Exploration, Preparation, Implementation and Sustainment factors related to how organizational and contextual variables affect adoption, implementation and early sustainability for provision of follow-up care, symptom, and risk management activities at 6 and 12 months post implementation. Aim 3 surveys 20 clinicians and staff members from 26 intervention practices (n=520) and conducts key informant interviews with 5 health care team members (who have participated in the survey; n=130) and 15 breast cancer survivors per practice (n=390; 5 per assessment point at baseline, 6 months and 12 months post intervention). Medical records of 20 patients with a history of breast cancer per practice per assessment point at baseline, 6 months and 12 months post intervention will be randomly selected for review (N=1,560) to assess and compare comprehensive breast cancer follow-up care outcomes. Sustainment will be measured through continued monitoring of the medical records for the 13 initial intervention practices at 18 and 24 months (N=520).

ELIGIBILITY:
Inclusion Criteria:

* Self-identification as a staff member or patient who has had breast cancer in a participating practice

Exclusion Criteria:

* Unable to speak, understand and/or read English
* Unable to provide informed consent

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 910 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Comprehensive Breast Cancer Follow-up Care | Repeated measures at baseline, 6 months, 12 months, 18 months and 24 months
  Percent of eligible recommendations performed per patient to assess the comprehensiveness of the follow up care received

CONTACTS AND LOCATIONS:
Overall Officials: Shawna V Hudson, PhD, Principal Investigator — Rutgers University
Locations (1):
- Rutgers University, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fadem SJ, Crabtree BF, O'Malley DM, Mikesell L, Ferrante JM, Toppmeyer DL, Ohman-Strickland PA, Hemler JR, Howard J, Bator A, April-Sanders A, Kurtzman R, Hudson SV. Adapting and implementing breast cancer follow-up in primary care: protocol for a mixed methods hybrid type 1 effectiveness-implementation cluster randomized study. BMC Prim Care. 2023 Nov 9;24(1):235. doi: 10.1186/s12875-023-02186-3. PMID 37946132